CLINICAL TRIAL: NCT02021292
Title: Prospective, Randomized, Placebo-controlled, Double-blind, Multicenter, Parallel-group, 24-week Study to Assess the Efficacy, Safety and Tolerability of Macitentan in Subjects With Inoperable Chronic Thromboembolic Pulmonary Hypertension
Brief Title: Clinical Study to Assess the Efficacy, Safety and Tolerability of Macitentan in Subjects With Inoperable Chronic Thromboembolic Pulmonary Hypertension
Acronym: MERIT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-055E201
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Chronic thromboembolic pulmonary hypertension (CTEPH)
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macitentan (Experimental): Macitentan 10 mg, oral tablet, to be taken once daily.
  Interventions: Drug: Macitentan
- Placebo (Placebo Comparator): Matching placebo oral tablet, to be taken once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Macitentan — Macitentan 10 mg, oral tablet, to be taken once daily.
  Other Names: ACT-064992
  Arms: Macitentan
Drug: Placebo — Matching placebo oral tablet, to be taken once daily.
  Arms: Placebo

SUMMARY:
Study to evaluate if macitentan is efficient, safe and tolerable enough to be used for treatment of inoperable chronic thromboembolic pulmonary hypertension (CTEPH).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Subject with CTEPH (WHO Group 4) judged as inoperable due to the localization of the obstruction being surgically inaccessible (i.e., distal disease).
* Female of childbearing potential must have a negative pre-treatment serum pregnancy test, be advised on appropriate methods of contraception, and agree to use 2 reliable methods of contraception.

Exclusion Criteria:

* Previous pulmonary endarterectomy.
* Recurrent thromboembolism despite sufficient oral anticoagulants.
* Symptomatic acute pulmonary embolism in the 6-month period prior to randomization.
* Known moderate-to-severe restrictive lung disease (i.e., TLC < 60% of predicted value) or obstructive lung disease (i.e., FEV1 < 70% of predicted, with FEV1/FVC < 65%) or known significant chronic lung disease diagnosed by chest imaging (e.g., interstitial lung disease, emphysema).
* Acute or chronic conditions (other than dyspnea) that limit the ability to comply with study requirements in the 3-month period prior to Screening visit or during the Screening period.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Papadakis, MD, Study Chair — Actelion
Locations (36):
- University Hospital Gasthuisberg / Interne Geneeskunde - I.G. Pneumologie, Leuven, Belgium
- China (6):
  - Beijing Chao-Yang Hospital-Department of Respiration, Beijing
  - Cardiovascular institute & Fuwai Hospital- Thrombus Center, Beijing
  - The first affiliated hospital of guangzhou medical university-respiratory department, Guangzhou
  - ngShanghai Pulmonary Hospital, Department of Pulmonary Circulation, Shanghai
  - The General Hospital of Shenyang Military Region,Congenital Heart Disease Department, Shenyang
  - Wuhan Asia Heart Hospital, Wuhan
- Centre for PPH, Charles University , II Interni klinika1.LF a VFN, Prague, Czechia
- France (3):
  - CHU de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Européen Georges Pompidou Service de Pneumologie, soins intensifs et endoscopies bronchiques, Paris
  - CHU de Toulouse Hopital Larrey, Toulouse
- Germany (3):
  - Justus-Liebig-Universität Gießen, Giessen
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Missionsärztliche Klinik gGmbH Akademisches Lehrkrankenhaus der Julius-Maximilians-Universität, Würzburg
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum, Kardiológiai Klinika, Debrecen
- Lietuvos Sveikatos Mokslų Universiteto Ligoninės Kauno Klinikos Pulmonologijos-Imunologijos Klinika, Kaunas, Lithuania
- Instituto Nacional de Cardiologia (INC) Ignacio Chavez, Mexico City, Mexico
- Poland (2):
  - Wojewódzki Szpital Specjalistyczny w Lublinie im. Stefana Kardynała Wyszyńskiego SPZOZ Oddział Kardiologii - Pododdział Intensywnego Nadzoru Kardiologicznego, Lublin
  - Wojewódzki Szpital Specjalistyczny we Wrocawiu, Wrocaw
- Russia (5):
  - Federal State Budgetary Institution "Scientific Research Institute of Systemic Problems of Cardiovascular Diseases", Siberian branch of RAMS, Kemerovo
  - Federal State Budgetary Institution "Russian Cardiology Scientific and Production Complex" of the Ministry of Health Care of the Russian Federation, Moscow
  - E.N.Meshalkin Novosibirsk State Research Institute Of Circulation Pathology Rosmedtechnology, Novosibirsk
  - Federal State Institution "Federal center of Heart, Blood and Endocrinology named after V.A.Almazov Rosmedtekhnologies", Saint Petersburg
  - Federal State Budgetary Institution "Research Institute for Cardiology" of Siberian Branch under the Russian Academy of Medical Sciences / Cardiovascular Surgery Department, Tomsk
- Severance Hospital, YonSei University Health System, Seoul, South Korea
- University Hospital Zürich, Zurich, Switzerland
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Division of Respiratory and Respiratory Critical Care Medicine, Bangkok
  - Siriraj Hospital, Division of Respiratory Disease and Tuberculosis, Bangkok
  - MAHARAJ NAKORN CHIANG MAI HOSPITAL, Department of Internal Medicine, Chiang Mai
- Istanbul University İstanbul Faculty Medicine Pulmonology Department, Capa_Istanbul, Turkey (Türkiye)
- Ukraine (2):
  - State Institute of Phthisiology and Pulmonology n.a. F.G. Yanovskiy of AMS Ukraine, Kyiv
  - Lviv Regional Clinical Hospital, Cardiosurgery Department, Lviv
- United Kingdom (3):
  - Papworth Hospital NHS Trust, Pulmonary Vascular Diseases Unit, Cambridge
  - Hammersmith Hospital, London
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Pulmonary Vascular Medicine, Sheffield

REFERENCES:
- [Result] Ghofrani HA, Simonneau G, D'Armini AM, Fedullo P, Howard LS, Jais X, Jenkins DP, Jing ZC, Madani MM, Martin N, Mayer E, Papadakis K, Richard D, Kim NH; MERIT study investigators. Macitentan for the treatment of inoperable chronic thromboembolic pulmonary hypertension (MERIT-1): results from the multicentre, phase 2, randomised, double-blind, placebo-controlled study. Lancet Respir Med. 2017 Oct;5(10):785-794. doi: 10.1016/S2213-2600(17)30305-3. Epub 2017 Sep 11. PMID 28919201
- [Derived] Kim NH, D'Armini AM, Howard LS, Jenkins DP, Jing ZC, Mayer E, Chamitava L, Lack G, Rofael H, Solonets M, Ghofrani HA. Long-Term Safety and Efficacy of Macitentan in Inoperable Chronic Thromboembolic Pulmonary Hypertension: Results from MERIT and its Open-Label Extension. Pulm Ther. 2025 Mar;11(1):101-116. doi: 10.1007/s41030-024-00276-w. Epub 2024 Nov 9. PMID 39520648
- [Derived] Ghofrani HA, Simonneau G, D'Armini AM, Fedullo P, Howard LS, Jais X, Jenkins DP, Jing ZC, Madani MM, Martin N, Mayer E, Papadakis K, Richard D, Kim NH; MERIT study investigators. Macitentan for the treatment of inoperable chronic thromboembolic pulmonary hypertension (MERIT-1): results from the multicentre, phase 2, randomised, double-blind, placebo-controlled study. Lancet Respir Med. 2024 Apr;12(4):e21-e30. doi: 10.1016/S2213-2600(24)00027-4. PMID 38548406

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 48 sites in 20 countries screened subjects for recruitment. The study was conducted (i.e., randomized subjects) in a total of 36 sites across 16 countries: Belgium, China, Czech Republic, France, Germany, Hungary, Lithuania, Mexico, Poland, Russia, Thailand, Turkey, South Korea, Switzerland, Ukraine, and the United Kingdom).
Pre-assignment Details: Target screening period from Visit 1 up to Randomization was maximum of 30 days, but longer period (up to 60 days) was permitted with pre-approval from Actelion. Total of 186 subjects were screened. Of these, 80 subjects were randomized in 1:1 ratio to macitentan 10 milligram (mg) (n = 40) and placebo (n = 40). All randomized subjects were treated.
Period: Overall Study
Arm/Group | Macitentan | Placebo
Started | 40 | 40
Completed | 40 | 37
Not Completed | 0 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macitentan | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 52
  >=65 years | 14 | 14 | 28
Age, Continuous [Median (Full Range); unit: years] | 60.0 [20 to 80] | 58.0 [23 to 78] | 59.0 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 14 | 15 | 29
Region of Enrollment [Count of Participants; unit: Participants] — Population: Asia includes: China, South Korea, Thailand; Eastern Europe: Czech Republic, Hungary, Lithuania, Poland, Russia, Ukraine; Latin America: Mexico; Western Europe: Belgium, France, Germany, Switzerland, Turkey and the United Kingdom.
  Participants
    Asia | 15 | 14 | 29
    Eastern Europe | 17 | 19 | 36
    Latin America | 1 | 1 | 2
    Western Europe | 7 | 6 | 13
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 25.7 [19.8 to 47.5] | 26.0 [18.3 to 36.2] | 25.7 [18.3 to 47.5]
Time since diagnosis of chronic thromboembolic pulmonary hypertension (CTEPH) [Mean (Standard Deviation); unit: years] | 1.7 (2.36) | 1.2 (1.95) | 1.5 (2.16)
6-minute walk distance (6MWD) [Mean (Standard Deviation); unit: meter] | 353.0 (87.90) | 351.2 (73.79) | 352.1 (80.64)
Pulmonary vascular resistance (PVR) [Mean (Standard Deviation); unit: dynes*sec/cm^5] | 929.2 (379.65) | 984.3 (487.06) | 956.8 (434.78)
WHO functional class [Count of Participants; unit: Participants] — Class I: no symptoms with exercise or at rest. Class II: No symptoms at rest but uncomfortable and short of breath with normal activity such as climbing a flight of stairs, grocery shopping, or making the bed. Class III: May not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting (e.g. doing normal chores around the house, have to take breaks while doing activities of daily living). Class IV: Symptoms at rest and severe symptoms with any activity. Most patients also have edema in the feet and ankles as result of right heart failure.
  Participants
    class I | 0 | 0 | 0
    class II | 12 | 6 | 18
    class III | 28 | 33 | 61
    class IV | 0 | 1 | 1
Use of pulmonary arterial hypertension (PAH) medication [Count of Participants; unit: Participants]
  NO | 16 | 15 | 31
  YES | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 16 in Pulmonary Vascular Resistance (PVR) at Rest.
Description: The primary efficacy endpoint is defined as the PVR at rest at Week 16 expressed as percent of baseline PVR at rest.
Time Frame: From baseline to Week 16
Population: Full analysis set included all subjects assigned to a study treatment.
Measure: Geometric Mean (95% Confidence Interval); unit: percent of baseline PVR
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 40 | 40
percent of baseline PVR | 73.0 [63.6 to 83.8] | 87.2 [78.5 to 96.7]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; The null hypothesis (change of PVR at rest in Week 16 in percent of baseline PVR in subjects treated with placebo or macitentan is the same) is tested on the primary endpoint by means of an analysis of covariance (ANCOVA) model on the log(e) transformed % of baseline PVR at rest at Week 16; Test type: Superiority; p = 0.0410, ANCOVA; ANCOVA model on log-transformed % of baseline PVR at Week 16 adjusted by treatment as a factor and log transformed PVR at baseline as a covariate; ratio of geometric means = 0.84, 95% CI 2-sided [0.70 to 0.99]

2. Secondary Outcome: Change From Baseline to Week 24 in Exercise Capacity, as Measured by the 6-minute Walk Distance (6MWD).
Description: The purpose of the six minute walk is to test exercise tolerance and capacity. The test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Time Frame: From baseline to Week 24
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 40 | 40
meter
  6MWD (m) at baseline | 353.0 (87.90) | 351.2 (73.79)
  6MWD (m) at Week 24 | 388.0 (83.31) | 352.2 (121.29)
  Change in 6MWD (m) from baseline to Week 24 | 35.0 (52.52) | 1.0 (83.24)
Statistical Analysis 1: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline in 6MWD at Week 24 is the same in the placebo and the macitentan group. Statistical model is ANCOVA including 6MWD at baseline as a covariate, with treatment as factor in the model; Test type: Superiority; p = 0.0326, ANCOVA — To control multiplicity across all endpoints, secondary endpoints were analyzed in sequence using hierarchical approach based on order and significance as pre-specified in protocol eliminating further adjustment for multiple comparisons; least squares (LS) mean difference = 34.04, 95% CI 2-sided [2.9 to 65.2]

3. Secondary Outcome: Change From Baseline to Week 24 in Borg Dyspnea Index Collected at the End of the 6-minute Walk Test (6MWT).
Description: This outcome measures the difference in the Borg dyspnea index collected at the end of the 6-minute walk test (6MWT) at Week 24 compared to baseline. The Borg dyspnea index rates the severity of dyspnea (difficult or labored breathing) on a scale from 0 ('Nothing at all') to 10 ('Very, very severe - maximal'). A decrease in the Borg dyspnea index indicates an improvement.
Time Frame: From baseline to Week 24
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 40 | 40
Score on a scale
  Borg dyspnea index score at baseline | 4.2 (2.52) | 4.2 (2.14)
  Borg dyspnea index score at Week 24 | 4.1 (2.52) | 4.4 (2.45)
  Change from baseline to Week 24 | -0.1 (1.86) | 0.3 (2.04)
Statistical Analysis 1: Comparison: Macitentan vs Placebo; The null hypothesis is that the mean change from baseline is the same in the placebo and the macitentan group. Statistical model is Analysis of Covariance including Borg dyspnea index at baseline as a covariate, with Treatment as factor in the model; Test type: Superiority; p = 0.3492, ANCOVA — [p-value comment as in outcome 2, analysis 1]; least squares (LS) mean difference = -0.39, 95% CI 2-sided [-1.21 to 0.43]

4. Secondary Outcome: Proportion of Subjects With Worsening in WHO Functional Class (FC) From Baseline to Week 24
Description: WHO functional classes are defined as follows: 1) class I: no symptoms with exercise or at rest. No limitation of activity. 2) class II: No symptoms at rest but slight limitation with ordinary activities causing symptoms (e.g. short of breath with climbing a flight of stairs, grocery shopping, or making the bed). 3) class III: may not have symptoms at rest but activities greatly limited by shortness of breath, fatigue, or near fainting. 4) class IV: symptoms at rest (such as dyspnea and/or fatigue) and inability to carry out any physical activity without symptoms (e.g. may faint especially while bending over with their heads lowered). Patients in class IV manifest signs of right heart failure. Shifting to a higher class (e.g. from class III to class IV) represents a 'worsening' while shifting to a lower class (e.g. from class III to class II) means an 'improvement'.
Time Frame: From baseline to Week 24
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 40 | 40
Participants
  WHO functional class I at baseline | 0 | 0
  WHO functional class II at baseline | 12 | 6
  WHO functional class III at baseline | 28 | 33
  WHO functional class IV at baseline | 0 | 1
  WHO functional class I at Week 24 | 3 | 1
  WHO functional class II at Week 24 | 15 | 10
  WHO functional class III at Week 24 | 22 | 26
  WHO functional class IV at Week 24 | 0 | 3
  Worsened | 0 | 3
  Not worsened - total | 40 | 37
  Not Worsened - unchanged | 31 | 29
  Not worsened - improved | 9 | 8
Statistical Analysis 1: Comparison: Macitentan vs Placebo; The null hypothesis is the odds of worsening are the same in the placebo and the macitentan group. Logistic regression is used for Treatment Group vs. Placebo comparison to generate odds ratio, confidence levels, and p-values with treatment and WHO functional class at baseline as factors in the model; Test type: Superiority; p = 0.0962, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.212, 95% CI 2-sided [0.001 to 1.464]

5. Post Hoc Outcome: Post-hoc Analysis of Change From Baseline to Week 16 in Pulmonary Vascular Resistance (PVR) at Rest Including Subjects With Corrected Hemodynamic Values
Description: The main analysis of the primary efficacy endpoint of PVR was repeated after the voluntary right heart catheterization source data verification (SDV) and independent medical review of hemodynamic data corrected for 13 subjects reported after the clinical database closure.
Time Frame: From baseline to Week 16
Population: Full analysis set for this post-hoc analysis included all subjects assigned to a study treatment with SDV values.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent of baseline PVR
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 40 | 40
Percent of baseline PVR | 71.5 [63.5 to 80.4] | 87.6 [79.0 to 97.2]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; The same statistical model as for the predefined analysis (ANCOVA) was applied, including 13 subjects with corrected hemodynamic values; Test type: Superiority; p = 0.0098, ANCOVA — This is the post-hoc analysis and p-value is an exploratory p-value; [statistical method as in outcome 1, analysis 1]; Model-adjusted geometric mean ratio = 0.81, 95% CI 2-sided [0.70 to 0.95]

6. Post Hoc Outcome: Post-hoc Analysis of Change From Baseline to Week 16 in Pulmonary Vascular Resistance (PVR) at Rest Excluding Subjects With Corrected Hemodynamic Values
Description: The main analysis of the primary efficacy endpoint of PVR was repeated which excluded data for 13 subjects with corrected hemodynamic values. The hemodynamic values were reported after the SDV assessment clinical database closure.
Time Frame: From baseline to Week 16
Population: Full analysis set excluding subjects with corrected hemodynamic values.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent of baseline PVR
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 33 | 34
Percent of baseline PVR | 68.4 [60.3 to 77.5] | 86.1 [77.3 to 95.7]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority; p = 0.0061, ANCOVA — This is the post-hoc analysis and p-value is an exploratory p-value; [statistical method as in outcome 1, analysis 1]; Model-adjusted geometric mean ratio = 0.79, 95% CI 2-sided [0.68 to 0.93]

7. Post Hoc Outcome: Post-hoc Analysis of Change From Baseline to Week 16 in Pulmonary Vascular Resistance (PVR) at Rest Excluding Subjects With Implausible Hemodynamic Findings
Description: The main analysis of the primary efficacy endpoint of PVR was repeated which excluded 14 subjects with implausible hemodynamic findings.
Time Frame: From baseline to Week 16
Population: Full analysis set excluding subjects with implausible hemodynamic findings.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent of baseline PVR
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 32 | 34
Percent of baseline PVR | 73.9 [66.2 to 82.4] | 86.6 [77.9 to 96.4]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority; p = 0.0414, ANCOVA — This is the post-hoc analysis and p-value is an exploratory p-value; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 0.85, 95% CI 2-sided [0.73 to 0.99]

8. Post Hoc Outcome: Post-hoc Analysis of Change From Baseline to Week 24 in Exercise Capacity, as Measured by the 6-minute Walk Distance (6MWD) Excluding Subjects With Implausible Hemodynamic Findings
Description: The same analysis for the secondary endpoint, 6MWD, is repeated on the full analysis set excluding 14 subjects with implausible hemodynamic findings.
Time Frame: From baseline to Week 24
Population: Full analysis set excluding subjects with implausible hemodynamic findings.
Measure: Least Squares Mean (95% Confidence Interval); unit: meter
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 32 | 34
meter | 37.41 [11.12 to 63.71] | 0.23 [-25.28 to 25.74]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority; p = 0.0468, ANCOVA — This is the post-hoc analysis and p-value is an exploratory p-value; Statistical model is ANCOVA including 6MWD at baseline as a covariate, with treatment as factor in the model; least squares (LS) mean difference = 37.19, 95% CI 2-sided [0.54 to 73.83]

ADVERSE EVENTS:
Time Frame: From double-blind study treatment initiation up to 30 days after study treatment discontinuation
Arm/Group | Macitentan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 2/40
Serious Adverse Events (participants affected / at risk) | 3/40 | 7/40
Other Adverse Events (participants affected / at risk) | 22/40 | 19/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=40) | Placebo (N=40)
Acute right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=40) | Placebo (N=40)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 6 (7) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4)
Oedema peripheral (General disorders) | 8 (10) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (3) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights.